CLINICAL TRIAL: NCT07259720
Title: Dento-Alveolar Changes in Maxillary Incisors After Orthodontic En-mass Retraction by Two Levels of Force Application
Brief Title: Dento-Alveolar Changes in Maxillary Incisors After En-Masse Retraction Using Two Power-Arm Heights
Acronym: DA-RET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Rania Alzany, Postgraduate Student - Orthodontics, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZH-ORTHO-RET-2025
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Malocclusion, Angle Class II, Division 1
Keywords: En-masse retraction Power arm lenghth CBCT Bone remodeling
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned into two parallel groups receiving different power-arm lengths (5 mm vs 9 mm) during en-masse retraction. Each group followed the same orthodontic protocol except for the intervention difference.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: 5 mm Power Arm (Experimental): Orthodontic en-masse retraction using temporary anchorage devices (TADs) with a 5 mm power arm height for force application. Maxillary incisors are retracted as a single unit following first premolar extraction.
  Interventions: Procedure: TAD-supported En-masse Retraction
- Group 2: 9 mm Power Arm (Experimental): Orthodontic en-masse retraction using temporary anchorage devices (TADs) with a 9 mm power arm height for force application. Maxillary incisors are retracted as a single unit following first premolar extraction.
  Interventions: Procedure: TAD-supported En-masse Retraction

INTERVENTIONS:
Procedure: TAD-supported En-masse Retraction — Orthodontic en-masse retraction of maxillary incisors using temporary anchorage devices (TADs) with different power arm heights following first premolar extraction. The intervention involves controlled retraction mechanics using a 0.017×0.025 stainless steel archwire and vertical power arms to alter the moment-arm and force system.

SUMMARY:
This study aims to evaluate the dento-alveolar changes associated with en-masse retraction of the maxillary anterior teeth using two different power-arm lengths to produce two distinct levels of force application. Twenty patients were randomly assigned into two equal groups. Group I received en-masse retraction using a 5-mm power arm, while Group II was treated using a 9-mm power arm. Cone-beam computed tomography (CBCT) was used to measure changes in buccal bone thickness at 3 mm, 6 mm, and 9 mm levels before and after retraction. The purpose of the study is to assess the influence of power-arm length on force direction, bone remodeling, and the safety of anterior tooth movement.

DETAILED DESCRIPTION:
The study was conducted to assess the dento-alveolar changes that occur during the en-masse retraction of maxillary anterior teeth when using two different power-arm lengths. Twenty orthodontic patients who required extraction of the maxillary first premolars as part of their treatment plan were included. Patients were selected according to well-defined inclusion criteria to ensure uniformity in skeletal pattern, dental status, and oral health. Any patients with previous orthodontic treatment, periodontal problems, or systemic conditions that could influence bone metabolism were excluded.

After obtaining approval from the Research Ethics Committee, participants were randomly divided into two equal groups. In Group I, retraction was carried out using a 5-mm power arm, while Group II was treated with a 9-mm power arm incorporated into the main archwire. All patients were treated with the same fixed orthodontic system, and temporary anchorage devices (TADs) were placed bilaterally to provide maximum anchorage. The archwire sequence, appointment intervals, and force application protocol were standardized for both groups to reduce variability.

Cone-beam computed tomography (CBCT) scans were taken for each patient before initiating retraction and after the completion of space closure. Buccal bone thickness was measured at three levels along the root (3 mm, 6 mm, and 9 mm from the cementoenamel junction). Measurements were recorded on the right and left sides and averaged. Additional clinical parameters-including the amount of anterior tooth movement, changes in incisor inclination, and any alterations in the occlusal plane-were evaluated to understand the mechanical implications of each power-arm length.

The main focus of the study was to determine how the length of the power arm affects the direction of force, the biomechanics of retraction, and the subsequent pattern of alveolar bone remodeling. All measurements were analyzed using appropriate statistical tests to compare differences between groups and between pre- and post-treatment values. The study aims to provide practical clinical guidance regarding the optimal choice of power-arm length to achieve effective, controlled anterior retraction while maintaining alveolar bone health.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged from 18 to 25 years. 2. Patients indicated for extraction of maxillary first premolars (those with Angle's Class I bimaxillary protrusion or Angle's Class II Division I malocclusion).

  3. Good oral hygiene. 4. Healthy compliant and motivated patient. 5. Full dentition in maxillary arch except wisdom teeth.

Exclusion Criteria:

* 1. Previous orthodontic treatments. 2. Any systemic or bone diseases. 3. Smoking history. 4. Presence of periodontal diseases.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Dentoalveolar changes of maxillary incisors after en-masse retraction using different power arm heights | Baseline (before retraction) and after space closure (approximately 6-9 months)
  Evaluation of maxillary incisor dentoalveolar changes following orthodontic en-masse retraction using temporary anchorage devices (TADs) with different power arm heights. Measurements include incisor inclination, root position, buccal and palatal alveolar bone thickness, and alveolar crest level changes assessed by CBCT.

CONTACTS AND LOCATIONS:
Locations (1):
- Orthodontic Department, Faculty of Dentistry - Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is retrospective and the data includes identifiable clinical and radiographic records that cannot be publicly released.

REFERENCES:
- See also: CBCT-based evaluation of en-masse retraction biomechanics. — https://pubmed.ncbi.nlm.nih.gov/35598724/